CLINICAL TRIAL: NCT04232228
Title: A UK Observational Study to Evaluate the Impact of Care4Today® IBD, a Smart System to Facilitate the Management of Crohn's Disease by Patients and Health Care Providers
Brief Title: A Study to Evaluate the Impact of Care4Today® IBD, a Smart System to Facilitate the Management of Crohn's Disease by Patients and Health Care Providers
Status: Terminated | Type: Observational
Why Stopped: The Care4Today® IBD dashboard for HCPs and the patient app will be deactivated indefinitely and will no longer be available for use
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108721; CNTO1275CRD4033 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Crohn's Disease (CD): Adult participants with moderate to severe CD who agree to be part of the study and who fit the inclusion/exclusion criteria and use Care4Today inflammatory bowel disease (C4T IBD) alongside standard of care (SOC) at participating centers will be observed. Data available per clinical practice and via the C4T IBD application will be collected within this study. Participants will also be asked to complete questionnaires that are sent directly to the patients, which are not completed as part of clinical practice or via the application. Relevant data will be collected by prospectively following participants from the index date for 12 months, and also by retrospectively collecting data for the 6-month period prior to the index date from participant's medical records. Index is the activation date of C4T IBD application in participant's smartphone.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was used in this study.

SUMMARY:
The purpose of this study is to describe the Crohn's Disease (CD)-related secondary healthcare resource utilisation of patients in the 6 months pre- and 12 months post-activation of Care4Today® inflammatory bowel disease (C4T IBD) alongside standard of care (SOC) in the management of CD.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe Crohn's disease (CD), diagnosed at least 6 months prior to index date, as documented by the treating healthcare professional (HCP)
* Participants with at least 6 months of continuous care in the study centre prior to index date
* Participants who have agreed to install Care4Today® inflammatory bowel disease (C4T IBD) on their iOS or android smartphone as part of their management of CD
* Participants providing informed written consent to participate in the study from the date of activation (including installation and linkage to HCP web interface) of the C4T IBD app on his/her smartphone

Exclusion Criteria:

* Participants with presence of ileorectal or ileal pouch-anal anastomosis documented in their medical records
* Participants in remission for over 2 years as documented in their medical records
* Participants participating in an interventional clinical trial
* Participants participating in an observational study where the protocol interferes with the C4T study in the opinion of the principal investigator at each site
* Participants with insufficient command of English to interact effectively with C4T IBD and complete the study questionnaires in the opinion of the principal investigator at each site
* Participants unable or unwilling to provide their informed written consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe CD for at least 6 months and with at least 6 months of continuous care, which may include conventional and/or biological therapies.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Crohn's Disease Related Secondary Health Related Utilization (HRU) in the 6 Months Pre-Activation of Care4Today® Inflammatory Bowel Disease (C4T IBD) Application (Pre-Index) | 6 months pre-index of C4T IBD application
  The number of gastroenterology health care provider (HCP) contacts per participant in the 6 months pre-index will be reported. Index is the activation date of C4T IBD application in participant's smartphone.
Crohn's Disease Related Secondary HRU in the 12 Months Post-Activation of C4T IBD Application (post-index) | Up to 12 months post index of C4T IBD application
  The number of gastroenterology HCP contacts per participant in the 12 months post-index will be reported. The 12 months post-index period will be split into two time periods: 0-6 months post-index and 6-12 months post-index. The 0-6 and 6-12 month post-index periods will be described separately.

SECONDARY OUTCOMES:
Crohn's Disease (CD)-Related Primary Healthcare Resource Utilization | 6 months pre- and 12-months post-index
  CD-related primary healthcare resource utilization of participants in the 6 months pre- and 12-months post-index of C4T IBD will be reported.
Number of Participants with Characteristics Including Duration of Disease, Current Treatments and Previous Treatments | At screening (during 6 months pre-index)
  Characteristics of participants enrolled into the study including, but not limited to, duration of disease, current treatments (ongoing at the time of C4T IBD activation) and previous treatments (including reasons for treatment changes where available) will be reported. Data will be collected from participant's medical records.
Disease Activity of Participants Measured Using the Harvey-Bradshaw Index (HBI) or Modified HBI | 6 months pre- and 12 months post-index
  Disease activity of participants using HBI or modified HBI will be reported.
Disease Activity of Participants Measured Using Markers of Systemic Inflammation | 6 months pre- and 12 months post-index
  Disease activity of participants using markers of systemic inflammation (Faecal calprotectin [FCP] and C reactive protein [CRP] levels) will be reported.
Disease Progression of Participants Measured Using the Fatigue Severity Scale (FSS) | Up to 12 months post-index
  FSS is a short questionnaire implemented in the C4T IBD application that allows a person to measure their level of fatigue. It contains 9 items measuring the severity of fatigue symptoms in the last week.
Disease Progression of Participants Measured Using Number of Bowel Movements | Up to 12 months post-index
  Number of daily bowel movements will be measured using the bespoke patient-reported outcome (PRO) within the C4T IBD application. The questionnaire captures bowel movements recorded as day/night, according to the level of urgency, and presence of blood.
Disease Progression of Participants Measured by Level of Abdominal Pain | Up to 12 months post-index
  Abdominal pain will be measured using the bespoke PRO within the C4T IBD application. The questionnaire captures the level of abdominal pain on a scale from 0-10 (at 2 points intervals) where higher score indicates more severe pain.
Impact of C4T IBD on Health Related Quality of Life (HRQoL, General and Inflammatory Bowel Disease [IBD] Specific) and Productivity | Up to 12 months post-index
  Impact of C4T IBD on HRQoL (general and IBD specific) and productivity will be reported based on online questionnaires.
Impact of C4T IBD on Participant's Level of Engagement with Their Disease Measured Using the Patient Activation Measure (PAM) | Up to 12 months post-index
  Impact of C4T IBD on participant's level of engagement with their disease measured using the PAM will be reported based on online questionnaire.
Patient- and HCP-Reported Satisfaction | Up to 12 months post-index
  Patient- and HCP-reported satisfaction of C4T IBD application will be reported based on bespoke online questionnaire.

OTHER OUTCOMES:
Change in Number of Flares | 6 months pre-index to 12 months post index
  Change in number of flares will be reported from 6 months pre-index to 12 months post index. Flares will be identified as recorded in medical notes. A flare is defined as an exacerbation of Crohn's disease.
Change in Duration of Flares | 6 months pre-index to 12 months post index
  Change in duration of flares will be reported from 6 months pre-index to 12 months post index. Flares will be identified as recorded in medical notes. A flare is defined as an exacerbation of Crohn's disease.
Change in Treatment Therapy | 6 months pre-index to 12 months post index
  Change in CD treatment therapy including steroid use will be reported.
Change in the Number of CD-Related Secondary HRU (Telephone calls, Outpatient Visits, Hospitalizations, Accident and Emergency Visits, Surgery) | 6 months pre- and 12-months post-index
  Change in the number of CD-related secondary HRU (telephone calls, outpatient visits, hospitalizations, accident and emergency visits and surgery) between the 6 months pre- versus 12 months post-activation of C4T IBD will be reported.
Change in the Number of CD-Related Primary HRU (Overall and by Type of HCP - General Practitioner [GP], Nurse) | 6 months pre- and 12-months post-index
  Change in the number of CD-related primary HRU (overall and by type of HCP - GP, nurse).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency